CLINICAL TRIAL: NCT01677338
Title: A Multi-center, Open-label Comparison Study of a 13C-uracil Breath Test Versus 99mTechnetium Sulfur Colloid Gastric Emptying Scintigraphy to Evaluate Normal, and Delayed Gastric Emptying Time in Dyspeptic Subjects
Brief Title: Phase 2 Study to Evaluate the Preliminary Performance of the C13-URA Breath Test Kit in Dyspeptic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: URA-12-001
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Dyspeptic Subjects
MeSH Terms: interventions — technetium Tc rhenium-sulfur colloid; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13C-uracil and 99mTc sulfur colloid (Experimental): Subjects will consume the Semi-solid Test Meal containing 500 uCi 99mTc sulfur colloid and 100 mg of 13C-uracil.
  Interventions: Drug: 13C-uracil; Drug: 99mTc sulfur colloid
- 99mTc sulfur colloid (Experimental): Subjects will consume the Solid Test Meal containing 500 uCi 99mTc sulfur colloid.
  Interventions: Drug: 99mTc sulfur colloid

INTERVENTIONS:
Drug: 13C-uracil — PO, the Semi-solid Test Meal containing 100 mg of 13C-uracil . Perform the Breath Test.
  Other Names: C13-URA
  Arms: 13C-uracil and 99mTc sulfur colloid
Drug: 99mTc sulfur colloid — PO, the Solid Test Meal containing 500 uCi 99mTc sulfur colloid. Perform the Scintigraphy.
  Other Names: Technetium Tc 99m Sulfur Colloid Injection

SUMMARY:
This study is a multi-center, open-label comparison study and aimed to evaluate the preliminary performance of this 13C-uracil GEBT to examine its abilities of identifying abnormal (delayed) gastric emptying rates in subjects.

DETAILED DESCRIPTION:
Approximately equal numbers of subjects will be enrolled in each of the 2 groups (with normal gastric emptying, and with delayed gastric emptying (gastroparesis)) to complete at least 10 subjects per group.

The subjects will first have their gastric emptying rates investigated by scintigraphy using the Solid Test Meal containing 500 uCi 99mTc sulfur colloid at Visit 1. Second, the subjects will have their gastric emptying rates investigated by scintigraphy and 13C-uracil GEBT simultaneously using the Semi solid Test Meal containing 500 uCi 99mTc sulfur colloid and 100 mg of 13C-uracil, respectively, at Visit 2. A comparison will be made between the results obtained at Visits 1 and 2 along with a comparison of the data obtained during Visit 2 for evaluation of the 13C-uracil GEBT.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [range is 18.0 to 33.0 kg/m2
* Subjects with any upper GI symptoms
* Stable creatinine

Exclusion Criteria:

* History of known peptic ulcers or stomach cancer.
* History of stomach surgery or resection
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food or other substance, unless approved by the investigator
* History of alcoholism or drug abuse
* History or presence of clinically significant GI, cardiovascular, central nervous system, hepatic, or renal disease; or other conditions
* History of eating disorders
* History or presence of an abnormal ECG, which, in the opinion of the investigator, is clinically significant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Expired 13CO2 concentrations | 6 hours
  Expired 13CO2 concentrations are obtained from breath test. The values will be calculated to Re(t)[B] semi-solid: remaining (%) of semi-solid test meal in stomach at t, t1/2[B] semi solid: half emptying time of semi-solid test meal , and tlag[B] semi-solid: lag time of semi-solid test meal.

SECONDARY OUTCOMES:
Concentrations of 13C-uracil and its major metabolites in plasma and urine | 6 hours
  PK parameters of 13C-uracil and its major metabolites, DHU and UPA, including AUCt, AUC∞, Cmax, tmax, λz, and t1/2,z, will be calculated based on plasma and urine concentration for 13C-uracil and its metabolites, and expired 13CO2-excretion, which calculated based on expired 13CO2 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Kimiyoshi Sudoh, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (2):
- United States (2):
  - Compass Research, Orlando, Florida
  - Dartmouth-Hitchcock Medical Center, Gastroenterology and Hepatology, Lebanon, New Hampshire